CLINICAL TRIAL: NCT06949631
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effects of Resistant Potato Starch on the Gut Microbiota Composition in Healthy Adults
Brief Title: Study on the Effects of Resistant Potato Starch on Gut Bacteria in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MSP Starch Products Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: M03-25-01-T0081
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Microbiota
Keywords: Gastrointestinal; Microbiota; Gut; healthy adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Potato Starch (Experimental): Active: 1 sachet per day oral
  Interventions: Dietary Supplement: Resistant Potato Starch
- Placebo (Placebo Comparator): Placebo: 1 Sachet per day oral
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resistant Potato Starch — Active Ingredients: 3.5 g potato starch Inactive ingredients: 3.5 g corn starch
  Arms: Resistant Potato Starch
Other: Placebo — Active Ingredients: N/A Inactive Ingredients: 7 g corn starch
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate how taking Resistant Potato Starch affects the gut microbiota compared to a placebo, in healthy adults. Over a 4-week period, participants will provide stool samples for analysis to detect any changes in gut bacteria. They will also record daily information in a diary about their stool consistency, frequency, digestive symptoms, and overall quality of life.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study designed to evaluate the effects of a low dose of Resistant Potato Starch on the gut microbiome in healthy adults. The test product is a type of resistant starch derived from potatoes, which may help strengthen the gut barrier and improve microbiome balance by acting as a prebiotic that supports healthy gut bacteria.

The main goal of the study is to measure changes in the gut microbiota after 4 weeks of taking the resistant starch compared to a placebo. Secondary goals include assessing changes in stool consistency, bowel movement frequency, digestive symptoms, and overall quality of life, also after 4 weeks of supplementation.

Before starting the study, participants will go through a short run-in period where they will complete a daily diary to track their stool form and frequency, general health changes, and any other medications they are taking.

The study will enroll generally healthy adults to specifically examine the effect of the resistant starch on levels of *Akkermansia*, a beneficial type of gut bacteria. People will be excluded from the study if they have taken the test product before, have a family history of gastrointestinal diseases, have used antibiotics within 5 weeks before or during the study, have existing gastrointestinal conditions, or have lactose and/or gluten intolerance. Anyone who, in the opinion of the Principal Investigator, may not be a good fit for the study or whose participation may pose a risk to their health will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Adults who are 18 to 69 years of age (inclusive).
2. Have a BMI between 18.0 to 34.9 kg/m2 (inclusive).
3. In good general health (i.e., no uncontrolled diseases or conditions) as deemed by the investigator, medical history, screening bloodwork, and are able to consume the study product.
4. Have maintained consistent dietary habits, including medication and supplement intake, and lifestyle for the last 3 months before screening and agree to maintain them throughout the study
5. Agree to follow the restrictions on concomitant treatments
6. Agree to follow the restrictions on lifestyle
7. Agree to use acceptable contraceptive methods
8. Willing and able to agree to the requirements of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study or demonstrate a positive pregnancy test at Visit 2.
2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
3. Individuals who have taken the TP at any time in the past, including having consumed products that list the TP as an ingredient.
4. Have a family history of peptic ulcer, colorectal cancer, or IBD.
5. Have structural or metabolic diseases/conditions that affect the GI system.
6. Presence of concomitant conditions such as organic GI disease, lactose and/or gluten intolerance, proneness to rectal bleeding due to hemorrhoids, or persistent GI problems (e.g., chronic constipation or diarrhea) which, in the opinion of the investigator, may interfere with study outcomes or participant safety.
7. Self-report of current or recovering acute GI problems at baseline (Visit 2).
8. Current diagnosis of IBS, dyspepsia, and/or significant GI disorders.
9. Screening alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP) results that are ≥ 2 times the upper limit of normal or any other clinically significant abnormal safety laboratory values as per the Investigator's discretion.
10. On an unstable dose of medication (i.e., less than 90 days at the same dose level)
11. Have Type I diabetes, uncontrolled Type II diabetes, uncontrolled high blood pressure (≥140 systolic or ≥90 diastolic mmHg), or uncontrolled thyroid disease ("uncontrolled" defined as being unmedicated, have an unstable use of medication within 3 months prior to screening, or have a stable use of medication for 3 months but still have uncontrolled conditions).
12. Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of the study product (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).
13. Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised (i.e., HIV/AIDS).
14. Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer), unless recovery occurred more than 5 years before the screening visit.
15. Are receiving treatments for or have been hospitalized in the last 12 months for psychiatric disorders (e.g., depression, bipolar disorder, schizophrenia, etc.).
16. Reports a clinically significant illness during the 28 days before the first dose of study product.
17. Major surgery in 3 months prior to screening or planned major surgery during the study.
18. Have a history of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program) or use that in the opinion of the investigator may be of a concern for the study.
19. Current enrollment or past participation in another study with any product(s) with at least one active ingredient within 28 days before screening or longer, if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
20. Any other medical condition/situation or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
To assess the shifts in Akkermansia genus in gut microbiota after 4 weeks of resistant potato starch (RPS) supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in the relative abundance of Akkermansia genus, as assessed via 16S ribosomal ribonucleic acid (rRNA) sequencing of fecal samples

SECONDARY OUTCOMES:
To assess the shifts in Bifidobacterium genus in gut microbiota after 4 weeks of RPS supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in the relative abundance of Bifidobacterium genus, as assessed via 16S rRNA sequencing of fecal samples
To assess the effect of RPS on stool form (consistency) after 3 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in consistency score and the incidence of the following stool types, as assessed by Bristol Stool Form Scale (BSFS) in daily diaries: Constipated stools (type 1 or 2)
To assess the effect of RPS on stool form (consistency) after 3 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in consistency score and the incidence of the following stool types, as assessed by Bristol Stool Form Scale (BSFS) in daily diaries:Diarrheal stools (type 6 or 7)
To assess the effect of RPS on the number of bowel movements (BM) (stool frequency) after 3 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in the average number of daily BMs, as assessed by daily diaries
To assess the effect of RPS on gastrointestinal (GI) symptoms after 4 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in GI symptoms, as assessed by Gastrointestinal Symptoms Rating Scale (GSRS)
To assess the effect of RPS on general well-being after 4 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in general well-being, as assessed by The World Health Organization Quality of Life - BREF (WHOQOL-BREF)
To assess the effect of RPS on health-related quality of life (QOL) after 4 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in health-related QOL, as assessed by RAND 36-Item Health Survey 1.0 (RAND-36)

OTHER OUTCOMES:
To assess the effect of RPS on leaky gut after 4 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in serum zonulin and lipopolysaccharide (LPS)
To assess the effect of RPS on systemic and gut microbial metabolomic biomarkers through metabolomic analyses of stool and serum samples after 4 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in abundance of gut microbiota and relevant metagenomic material, identified in metagenomic analyses of stool samples
To assess the effect of RPS on gut microbiota composition and determine the underlying genetic mechanisms through metagenomic analyses of stool samples after 4 weeks of supplementation, compared to a placebo | Week 4
  Change from baseline to Week 4 in abundance of gut microbiota and relevant metagenomic material, identified in metagenomic analyses of stool samples
To assess the safety of RPS | From Week 1 to Week 4
  Reports of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bush, Chief Scientific Officer, Study Director — MSP Starch Products Inc.
Locations (1):
- Apex Trials, Guelph, Ontario/ON, Canada

IPD SHARING:
Plan to Share IPD: No